CLINICAL TRIAL: NCT06068322
Title: Effects and Mechanisms of Supramaximal High-Intensity Interval Training in People With and Without Chronic Obstructive Pulmonary Disease on Extrapulmonary Manifestations
Brief Title: Supramaximal High-Intensity Interval Training in People With and Without Chronic Obstructive Pulmonary Disease
Acronym: COPD-HIIT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Umeå University (Other)
Collaborators: Hasselt University (Other); Swedish Heart Lung Foundation (Other); European Research Council (Other); The Swedish Research Council (Other Government); Ziekenhuis Oost-Limburg (Other); Strategic Research Area - Health Care Science (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: COPD-HIIT RCT; 2020-01296 (Other Grant/Funding Number: The Swedish Research Council); 2020-0139 (Other Grant/Funding Number: The Swedish Heart-Lung Foundation); 101078602 (Other Grant/Funding Number: The European Research Council)
Record Dates: First submitted 2023-06-26; First posted 2023-10-05 (Actual); Last update posted 2024-05-23 (Actual); Status verified 2024-05

CONDITIONS: COPD; Healthy Controls
Keywords: Chronic obstructive Pulmonary Disease; Pulmonary Disease, Chronic Obstructive; Chronic airway disease; COPD; physical activity; exercise
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Motor Activity

STUDY DESIGN:
Intervention Model Description: In Phase 1, participants will be randomised to either interventional arm or control arm with a 1:1 allocation ratio, using a computer-generated block randomisation schedule stratified for sex (male, female), age and centre with equal allocation to all study arms. For Phase 2 only the participants with COPD will continue the maintenance program in their allocated group. A usual of care group consisting of patients with COPD will also be recruited to serve as control in the maintenance part.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The outcome assessors and data analysts will be masked to group allocation. The participants will be given repeated instructions not to reveal their group allocation to the outcome assessors. The dataset will be blinded regarding group allocation when performing analyses.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Supramaximal high-intensity interval training (Supramaximal HIIT) (Experimental): Each HIIT session consists of 10 repeated 6-seconds regulated high intensity cycling sprints against an individualized load set to reach a supramaximal exercise intensity (i.e. power output is higher than power output at maximum oxygen uptake). Session duration for HIIT is initially 20 min, including warm-up (5 min) and cool-down (5 min). The protocol enables controlled and systematic adjustments of training intensity by means of standardized criteria.
  Interventions: Other: Exercise training on a stationary bicycle
- Moderate-intensity continuous training (MICT) (Active Comparator): Each MICT session will consist of aerobic training regulated against an individualized load set to reach a moderate submaximal exercise intensity (i.e. power output is lower than power output at maximum oxygen uptake). Session duration for MICT is initially 30 min, including warm-up (5 min) and cool-down (5 min). The protocol enables controlled and systematic adjustments of training intensity by means of standardized criteria.
  Interventions: Other: Exercise training on a stationary bicycle
- Usual care (No Intervention): The passive control group will receive usual care alone and a standardized phone call every three months including assessments of health status (CAT), disease specific quality of life (CRQ) and questions on symptoms of exacerbations. We will match the participants in the standard care group to those randomized to HIIT or MICT by age, sex, disease severity, educational level, and physical activity.

INTERVENTIONS:
Other: Exercise training on a stationary bicycle — Training is performed two to three times per week for a total of 30 sessions using a group format.
  Both regimens start with a five-minute warm-up and ends with a five-minute cool-down, performed at an intensity corresponding to 30% of the maximal work rate achieved during a CPET (i.e., max aerobic power [MAP]) with a self-selected pedalling cadence of 50-70 revolutions per minute (RPM).
  All exercise sessions will be held and supervised by an experienced health care professional, i.e. physiotherapists or other health professional.
  The different types of exercise training is described under the specific arm.
  Following the first 12-week training period, participants with COPD will enter a 21-month maintenance phase. They will continue to exercise using the same training modality (HIIT or MICT) as during the first 12-weeks but can select between three different settings to continue their training: "Home", "Outpatient", or "Mix" setting.
  Arms: Moderate-intensity continuous training (MICT); Supramaximal high-intensity interval training (Supramaximal HIIT)

SUMMARY:
Beyond pulmonary complications, COPD presents with extrapulmonary manifestations including reduced cognitive, cardiovascular, and muscle function. While exercise training is the cornerstone in the non-pharmacological treatment of COPD, there is a need for new exercise training methods.

The COPD-HIIT trial intend to investigate the effects and mechanisms of 12 weeks supramaximal high-intensity interval-training (HIIT) compared to moderate intensive continous training (MICT) in people with COPD and matched healthy controls on important clinical outcomes.

The trial also intends to compare the effects of 24 months of exercise training (supramaximal HIIT or MICT) to usual care in people with COPD on brain health, cardiorespiratory fitness and muscle power; in people with COPD.

DETAILED DESCRIPTION:
COPD-HIIT is a prospective, multi-centre, randomised, controlled, parallel-group superiority trial with assessor and data analyst blinding, featuring a 1:1 allocation ratio and two separate phases. In Phase 1, the trial will investigate the effects and mechanisms of a 12 week intervention with supramaximal HIIT compared to MICT in people with COPD and matched healthy controls. Upon completing the initial 12 week intervention and follow-up assessments, people with COPD, but not healthy controls, will enter Phase 2 of the trial. Phase 2 comprises a 21 month maintenance exercise program. Subsequently, exercise training (supramaximal HIIT or MICT) will be performed until a 24 month follow-up. A separate control group of people with COPD, receiving usual care only, will undergo assessments at baseline and 24-months, making Phase 2 a partially randomized controlled trial.

The primary objectives are:

1. to determine and compare the effect of 12-weeks of supramaximal HIIT and MICT on cognitive function, cardiorespiratory fitness, and muscle power in people with COPD compared to matched healthy controls (Phase 1).
2. to determine and compare the effect of 24-months of supramaximal HIIT, MICT and usual care on cognitive function, cardiorespiratory fitness and muscle power in people with COPD (Phase 2).

Phase 1 and 2 of the COPD-HIIT project will be performed at two recruiting centres. 1) Department of Community Medicine and Rehabilitation, Physiotherapy, Umeå University, Umeå, Sweden and Norrlands Universitetssjukhus, and 2) Faculty of Rehabilitation Sciences, Hasselt University, Diepenbeek, Belgium and Ziekenhuis Oost-Limburg (ZOL, Genk, Belgium).

In Phase 1, eligible participants will be randomized to either supramaximal HIIT (intervention arm) or MICT (active control arm) on a stationary bicycle (Smart ZBike, Zycle, Valencia, Spain). For both arms, training is performed two to three times per week for a total of 30 sessions (Table 1) using a group format with groups of 4-8 participants at the same time. Both protocols enable controlled and systematic adjustments of training intensity by means of standardized criteria to achieve a progressive overload

Regarding supramaximal HIIT, importantly, while the intensity is supramaximal, it is dosed and performed at a given fraction of the maximum capacity that the person can produce during the bout (6-seconds). In contrast to an all-out regimen, or sprint interval training (SIT), this allows for the introduction and titration of intensity to the highest acceptable level without the individual feeling unwell during the process.

In Phase 2, participants with COPD will enter a 21 month maintenance phase. They will continue to exercise using the same training modality (HIIT or MICT) as during the first 12-weeks but can select between three different settings to continue their training: "Home", "Outpatient", or "Mix" setting. Notably, the participant can, at any time during the maintenance period, change between the "Home", "Outpatient" or "Mix" settings when conducting their endurance training. Irrespective of the originally assigned group (supramaximal HIIT or MICT) or if the participant selects to continue in "Home", "Outpatient" or "Mix" setting, they will also perform a resistance training (RT) regime. The RT regime will consist of ten lower and upper-body exercises designed following American College of Sports Medicine guidelines and other relevant RT literature for increasing muscular strength, endurance, and power.

All exercise sessions will be held and supervised by an experienced health care professional, such as physiotherapists, exercise physiologists or other health professional with equivalent expertise. All intervention providers will receive training on exercise intervention protocols to ensure standardization among centres.

The between-group effects will be analyzed using analysis of covariance (ANCOVA). In the ANCOVA, baseline values, age, sex, center and VO2peak will be used as covariates. There will be one model for the COPD group and one for HC. To investigate any differential effects to the interventions between COPD and HC, an additional model including the Group (COPD/HC) × Intervention (HIIT/MICT) will be performed. Furthermore, pre-specified longitudinal mediation analyses will be performed on the entire MRI and PET/CT sample between changes in VO2peak, neurodegenerative measures, e.g., cognitive function and hippocampal volume, and inflammation levels between baseline and 24 months.

Analyses will employ the intention-to-treat when applicable. Meaning that all participants randomized, whether they receive their allocated intervention or withdrew from the trial, will be included in the analysis. The primary analyses are performed using Multiple Imputation by Chained Equations (MICE) for missing data. The imputation will be done separately for each intervention arm. In addition, a per-protocol analysis (defined as > 75% attendance rate as well as no exacerbations during the last two weeks prior to follow-up assessment), and a complete-case analysis (including participants with complete outcome measurements independent on attendance rate) will be reported.

The full study protocol adheres to the SPIRIT guidelines and its outcomes extension, with intervention descriptions further guided by the TIDieR checklist the Consensus on Exercise Reporting Template (CERT). Publications from COPD-HIIT will follow the CONSORT statement, or relevant guidelines at the time of publication. Publications including qualitative outcomes will also be guided by the Consolidated Criteria for Reporting Qualitative Research (COREQ).

ELIGIBILITY:
The inclusion criteria are:

1. 60 years of age or older
2. Independent in activities of daily living
3. For people with COPD: Symptomatic (COPD assessment test [CAT] ≥10 or modified Medical Research Council dyspnea scale [mMRC] ≥2) or not being regularly physically active at a moderate or high intensity over the last year defined as not meeting WHO requirements for physical activity.
4. For people with COPD: Post-bronchodilator spirometry confirmed COPD diagnosis (forced expiratory volume in one second (FEV1) to forced vital capacity (FVC) ratio < 0.70).
5. For healthy controls: Normal lung function

The exclusion criteria are:

1. Movement related conditions, cardiovascular, neuromuscular, metabolic, skeletal and/or rheumatic conditions and diseases that are unstable and/or prohibits exercise or tests, based on screening by a physician. For example, but not limited to:

   I. Musculoskeletal pain prohibiting participation in tests and exercise II. Recent myocardial infarction, coronary artery bypass grafting, angioplasty, or other cardiac events III. Uncontrolled arterial hypertension IV. Pathological ECG-findings during CPET
2. Other lung conditions, including, but not limited to asthma, interstitial lung disease, lung cancer, pulmonary hypertension, pulmonary vascular disease, pulmonary fibrosis
3. Medical conditions and treatments with known effects on brain function and cognition, for example:

   I. Previous trauma to the head with lasting cognitive or symptom-related issues II. Physical or mental disabilities III. Neurological condition (dementia, multiple sclerosis, stroke) IV. Psychiatric illness, not including depression or general anxiety disorder V. Severe cognitive impairment VI. Recent or current cancer diagnosis and treatment
4. For those accepting MRI or PET/CT: metal implants, pacemakers, claustrophobia and other MRI incompatible factors.
5. Inability to read or speak Swedish (Umeå participants), Dutch, French (Hasselt participants) or English (Umeå and Hasselt participants).
6. For people with COPD:

I. Co-morbid conditions that limit exercise performance to a greater extent than the COPD diagnosis.

II. Currently participating in a pulmonary rehabilitation program or have been involved in pulmonary rehabilitation in the last 12 months.

III. Experienced a COPD exacerbation that led to a change in medication dosage or frequency in the preceding six weeks.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 208 (Estimated)
Dates: Start 2023-11-09 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline global cognitive function | Baseline, 12 weeks, 24 months
  Global cognitive function will be assessed as the Z-score determined by the combined performances on six tests from the Cambridge Neuropsychological Test Automated Battery (CANTAB) and the trail making test (TMT-A, TMT-B). The following tests from the CANTAB will be used: Motor screening task, reaction time, visual information processing, paired associates learning, spatial working memory, verbal recognition memory. The test battery takes around 60 minutes to complete. The test scores from the seven tests will be combined into a composite Z-score. The Z-score describes how much a point deviates from a mean or specific point. The Z-score represents how many standard deviations an individual's score is from the mean score of the reference population, which is represented as zero.
Change from baseline cardiorespiratory fitness | Baseline, 12 weeks, 24 months
  Measured as maximum oxygen uptake (VO2peak [ml O2/min/kg]) during a standardized ramp-protocol cardiopulmonary exercise test (CPET) on a cycle ergometer. The CPET will start with a 3-minute resting phase before a 3-minute unloaded (or lowest wattage possible) warm-up phase. The aim is to have a ramp-phase of 8-12 minutes, until the participant stops due to voluntarily exhaustion, symptom-limitation or failure to maintain a cadence of 50-70 RPM.
Change from baseline quadriceps muscle power | Baseline, 12 weeks, 24 months
  Peak power (Nm/s) assessed during a seated leg extension in a dymanometer (Biodex System 4). Participants will be instructed to extend their leg as fast and as hard as possible and then passively return the leg to the starting position.

SECONDARY OUTCOMES:
Change from baseline brain structure | Baseline, 12 weeks, 24 months
  Assessed using standard MRI-sequences including in a 3 Tesla MRI-scanner. T1-weighted images will be used to determine volumes of grey matter, white matter and lateral ventricle size. T2-weighted, fluid-attenuated inversion recovery (FLAIR), and susceptibility weighted (SW) images are collected to assess perivascular spaces, lacunes, white-matter lesions and microbleeds. For structural MRI data volume (mm3), area (mm2) and cortical thickness (mm) will be the unit of measure.
Change from baseline brain activity | Baseline, 12 weeks, 24 months
  Task-based functional MRI will be performed to evaluate brain activity in the hippocampus and prefrontal cortex, measured as BOLD signal change.The face-name association task will be used.
Change from baseline cerebral perfusion | Baseline, 12 weeks, 24 months
  Assessed using arterial spin labelling (ASL) in a 3T MRI-scanner (mL/100g/minute).
Change from baseline neuroinflammation | Baseline, 12 weeks, 24 months
  In vivo neuroinflammation is measured as uptake rate (ki) of 11C-deprenyl in the brain assessed with PET/CT (General Electric, WI, USA) under resting-state conditions after intravenous injection of 314 MBq of 11C-Deprenyl. . Uptake rate of 11C-deprenyl in the brain is modeled with Patlak analyses, where higher uptake is representative of higher levels of inflammation.
Change from baseline exercise tolerance | Baseline, 12 weeks, 24 months
  Test duration (mm:ss) on a constant-workload cycle test (CWRT) set at 75% of maximal power achieved during a CPET. After a 3-minute resting phase and a 3-minute warm-up phase at 30% of MAP, participants will cycle at a constant workload corresponding to 75% of MAP with a self-selected pedaling cadence of 50-70 RPM. Participants will be instructed to exercise for as long as possible.
Change from cardiorespiratory fitness | Baseline, 6 weeks
  A intermediate test at 6-weeks will be done to regulate training intensity and the result will be used as a secondary outcome. Measured as maximum oxygen uptake (VO2peak [ml O2/min/kg]) during a standardized ramp-protocol cardiopulmonary exercise test (CPET) on a cycle ergometer. The CPET will start with a 3-minute resting phase before a 3-minute unloaded (or lowest wattage possible) warm-up phase. The aim is to have a ramp-phase of 8-12 minutes, until the participant stops due to voluntarily exhaustion, symptom-limitation or failure to maintain a cadence of 50-70 RPM.
Change from baseline lactate concentration during constant-workload cycle test (CWRT) | Baseline, 6 weeks, 12 weeks, 24 months
  Capillary blood lactate (mmol/L) will be measured during and immediately after the CWRT to assess the metabolic demand.
Change from baseline cognitive function: Motor screening task | Baseline, 12 weeks, 24 months
  Test score in the CANTAB Motor screen task. During the test, colored crosses appear in different locations on the screen. The participant must select the cross as quickly and accurately as possible.
Change from baseline cognitive function: Reaction time | Baseline, 12 weeks, 24 months
  Test score in the CANTAB reaction time test. During the test, participants must select a button on the screen. Circles are presented above the button and the participant is asked to react as soon as possible once a yellow dot appears in one of the circles by clicking the corresponding circle.
Change from baseline cognitive function: Visual information processing | Baseline, 12 weeks, 24 months
  Test score in the CANTAB Visual information processing test. During the test, a white box is shown in the center of the screen where digits from 2 to 9 appear in a pseudo-random order at the rate of 100 digits per minute. Participants are requested to detect target sequences of digits (e.g., 2-4-6, 3-5-7, 4-6-8). When the participant sees the target sequence, they must respond by selecting the button in the center of the screen as quickly as possible.
Change from baseline cognitive function: Paired associates learning | Baseline, 12 weeks, 24 months
  Test score in the CANTAB Paired associates learning test. In the test, boxes are displayed on the screen and are opened in a randomized order. One or more of them will contain a pattern. The patterns are then displayed in the middle of the screen, one at a time and the participant must select the box in which the pattern was originally located.
Change from baseline cognitive function: Spatial working memory | Baseline, 12 weeks, 24 months
  Test score in the CANTAB spatial working memory test. During the test, several colored boxes are shown on the screen. The aim of this test is that, by selecting the boxes and using a process of elimination, the participant should find one yellow 'token' in each of several boxes and use them to fill up an empty column on the right-hand side of the screen
Change from baseline cognitive function: Executive function | Baseline, 12 weeks, 24 months
  Test score in the trail making test. The TMT consists of two parts, A and B and is performed with paper and pencil. During part A, the participant needs to connect 25 digits in ascending order as fast as possible by drawing lines between the digits. During part B, the participants need to connect 13 digits in ascending order and 12 letters in alphabetical order, alternating digits, and letters (i.e., 1 - A - 2 - B - 3 - C, etcetera) as fast as possible by drawing lines between the digits and letters.
Change from baseline anaerobic exercise capacity | Baseline, 12 weeks, 24 months
  Intensity (produced power, in watts) at the final stage during a Borg cycle strength test (BCST). The BCST is a submaximal cycle ergometer test that is used to estimate maximum mean power output for 30 seconds (MPO30) without an all-out effort. The BCST consists of 30-second efforts with increasing intensity, interspersed with 30-seconds passive recovery between each effort. With a target pedaling cadence of 80-90 RPM, participants cycle until they score an RPE of ≥17, or when they cannot keep the target cadence (<75 RPM for five seconds).
Change from baseline cognitive function: Verbal recognition memory | Baseline, 12 weeks, 24 months
  Test score in the CANTAB verbal recognition memory test. During the test, the participant is shown a list of words to remember. During the recognition phase, the participant is asked to say whether they remember seeing the word on the screen before. The word can be one of the originals, or a new word (distractor) which they have not yet seen before.
Change from baseline chronic inflammation | Baseline, 12 weeks, 24 months
  Levels of hs-CRP in venous blood. Unit of measure is mg/L.
Change from baseline inflammatory markers | Baseline, 12 weeks, 24 months
  Llevels of interleukin-6, interleukin-8 and TNF-alpha in venous blood. Unit of measure is pq/mL.
Change from baseline fibrinogen | Baseline, 12 weeks, 24 months
  Plasma levels of fibrinogen. Unit of measure is g/L.
Change from baseline blood cell count | Baseline, 12 weeks, 24 months
  White blood cells and eosinophils measured in whole blood. Unit of measure is count x 10^9/L.
Change from baseline neurotrophic factors | Baseline, 12 weeks, 24 months
  Levels of BDNF, irisin, IGF-1, Cathepsin B and clusterin in venous blood samples. Unit of measure is pq/ml.
Change from baseline resting lactate | Baseline, 12 weeks, 24 months
  Concentration of lactate in capillary blood samples. Unit of measure is mmol/L.
Change from baseline blood lipid profile | Baseline, 12 weeks, 24-months
  Total cholesterol, LDL, HDL, non-HDL and triglycerides. Unit of measure is mmol/L.
Change from baseline metabolic function: Glucose | Baseline, 12 weeks, 24-months
  Plasma levels of glucose in fasted venous blood sample. Unit of measure is mmol/L.
Change from baseline metabolic function: Insulin | Baseline, 12 weeks, 24-months
  Plasma levels of insulin in fasted venous blood sample. Unit of measure is mIU/L.
Change from baseline metabolic function: Insulin resistance | Baseline, 12 weeks, 24-months
  Levels of glucose and insulin levels will be used to calculate the HOMA-IR (Homeostatic Model Assessment of Insulin Resistance). The unit of measure is arbitrary units where values above 1.9 indicates early insulin resistance, and above 2.9 indicates significant insulin resistance.
Change from baseline metabolic function: Glycated hemoglobin | Baseline, 12 weeks, 24-months
  Levels of Hb1Ac, measured as a percentage (%) of red blood cells that is bound to glucose.
Change from baseline quadriceps muscle strength | Baseline, 12 weeks, 24 months
  Muscle strength will be determined as the one-repetition maximum (1-RM) defined as the maximum torque (Nm/s) able to be lifted through the full range of motion during seated leg extension in the dominant leg, using a dymanometer (Biodex System 4)
Change from baseline quadriceps muscle endurance | Baseline, 12 weeks, 24 months
  Defined as the maximum number of repetitions able to be lifted with a good technique through the full ROM at an intensity corresponding to 45% of 1-RM, during seated leg extension in the dominant leg, using a dymanometer (Biodex System 4).
Change from baseline functional performance: Five time sit-to-stand test (5-STS) | Baseline, 12 weeks, 24 months
  Time needed (in seconds) to complete the 5-STS.
Change from baseline functional performance: Stair climbing power test | Baseline, 12 weeks, 24 months
  Time needed (in seconds) to ascent a 10-step flight of stairs.
Change from baseline muscle fibre size | Baseline, 12 weeks
  The tissue sample obtained from the vastus lateralis muscle will be examined with morphometric analyses to determine cross-sectional fiber area of all fibres and per subtype. Unit of measurement is square micrometers.
Change from baseline proportion of slow and fast subtypes of contractile myosin heavy chain isoforms | Baseline, 12 weeks
  The tissue sample obtained from the vastus lateralis muscle will be examined with immunohistochemistry techniques to categorize fiber types. Expressed as relative distribution in percent and relative area of the muscle in percent.
Change from baseline capillary density | Baseline, 12 weeks
  The tissue sample obtained from the vastus lateralis muscle will be examined with morphometric analysis to determine capillary density, estimated as the total number of capillaries per millimeter squared muscle cross-section.
Change from baseline capillaries per fiber | Baseline, 12 weeks
  The tissue sample obtained from the vastus lateralis muscle will be examined with morphometric analysis to determine the number of capillaries in close contact with each muscle fiber. Unit of measure is number of capillaries in close contact with fibre.
Change from baseline capillaries to fiber area | Baseline, 12 weeks
  The tissue sample obtained from the vastus lateralis muscle will be examined with morphometric analysis to determine the number of capillaries around each fiber relative to its cross-sectional area.
Change from baseline capillaries sharing factor | Baseline, 12 weeks
  The tissue sample obtained from the vastus lateralis muscle will be examined with morphometric analysis to determine the capillary-to-fiber ratio
Change from baseline myofiber and mitochondrial disruption/abnormalities (NADH-TR) | Baseline, 12 weeks
  Staining of reduced nicotinamide adenine dinucleotide-tetrazolium reductase, succinate dehydrogenase, and cytochrome c oxidase. Measured as % of fibers with abnormal staining pattern and fiber area in µm2 of fibers with abnormal staining pattern.
Change from baseline mitochondrial biogenesis | Baseline, 12 weeks
  mRNA and protein levels of peroxisome proliferator-activated receptor gamma coactivator 1 (PGC-1) alpha and PGC-1beta. Unit of measure is fold-change or arbitrary units.
Change from baseline enzyme activity | Baseline, 12 weeks
  Enzyme activities of phosphofructokinase (PFK; glycolysis), lactate dehydrogenase (LDH; anaerobic glycolysis), citrate synthase (CSM Krebs cycle), succinate dehydrogenase (SDH; Krebs cycle), 3-hydroxyacyl Coenzyme A dehydrogenase (HADH; beta-oxidation) and mitochondrial complex I-V. Unit of measure is micromol/min/g tissue.
Change from baseline enzyme content | Baseline, 12 weeks
  Enzyme content of phosphofructokinase (PFK; glycolysis), lactate dehydrogenase (LDH; anaerobic glycolysis), citrate synthase (CS; Krebs cycle), succinate dehydrogenase (SDH; Krebs cycle), 3-hydroxyacyl Coenzyme A dehydrogenase (HADH; beta-oxidation) and mitochondrial complex I-V. Unit of measure is micromol/min/g tissue.
Change from baseline angiogenesis | Baseline, 12 weeks
  mRNA and protein level of VEGF (fold change or arbitrary units).
Change from baseline proteins related to muscle-brain cross talk | Baseline, 12 weeks
  mRNA and protein level of BDNF, fibronectin type III domain-containing protein 5 (FNDC5) and kynurenine aminotransferase (KAT1-4). Unit of measure is fold change and arbitrary units.
Change from baseline modulation of autonomic cardic function | Baseline, 12 weeks, 24 months
  Resting heart rate variability measured in the time domain as the root mean square of the successive differences (RMSSD, in milliseconds), and time domain (LH:HF ratio) using a chest strap heart rate monitor.
Change from baseline blood pressure | Baseline, 12 weeks, 24 months
  Resting blood pressure, measured as systolic and diastolic pressure in mmHg.
Change from baseline epigenetic modifications in muscle samples | Baseline, 12 weeks
  Samples will be analysed for genome-wide DNA methylation, via the EPICarray technology.
Change from baseline epigenetic modifications in blood samples | Baseline, 12 weeks, 24 months
  Whole blood EDTA samples will be analysed for genome-wide DNA methylation, via the EPICarray technology.
Change from baseline body composition | Baseline, 12 weeks, 24 months
  Body composition measures include body mass index, waist and hip circumference (cm), percentage of body fat, fat-free mass (kg), and fat-free mass index (kg/m2). Fatmass and fatfree mass is measured with bioelectrical impedance.
Change from baseline impact of COPD in daily life | Baseline, 12 weeks, 6 months, 12 months, 15 months, 18 months, 21 months and 24 months
  Measured vid the COPD Assessment Test (CAT)
Change from baseline disease specific quality of life | Baseline, 12 weeks, 6 months, 12 months, 15 months, 18 months, 21 months and 24 months
  Measured with the chronic respiratory disease questionnaire (COPD group only). The CRQ measures the impact of chronic respiratory disease on HRQoL and covers four key domains of HRQoL, including: dyspnea, fatigue, emotional function, and mastery. Each item is scored on a 7-point Likert scale; scores within each domain are summated for a total score per domain.
Change from baseline Health related quality of life | Baseline, 12 weeks, 24 months
  Measured with the EQ-5D-5L questionnaire.It assesses an individual's HRQoL in five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression91. Each dimension has five response levels, ranging from level 1 (no problems) to level 5 (extreme problems). By combining one level from each dimension, a health state ranging from 11111 (the best health state) to 55555 (the worst health state) is defined and converted into an index score using a scoring algorithm.
Change from baseline state of depression and anxiety | Baseline, 12 weeks, 24 months
  The Hospital Anxiety and Depression Scale (HADS) will be used to assess states of depression and anxiety. The HADS is a reliable 14-item questionnaire regarding feeling of depression and anxiety in the past week which can be answered within 2 - 5 minutes. A separate score is given for depression and anxiety. where a higher score means higher severity.
Self-percieved change | 12 weeks, 24-months
  Self-perceived change in outcomes will be measured via the Global Rate of Change scale with the purpose to quantify the extent to which a participant's outcomes have improved or deteriorated over time. Participants will provide an answer via a 11-point Likert scale (-5 = "Much worse"; 0 = "Unchanged"; 5 = "Much better").
Number of responders | 12 weeks, 24-months
  Total amount of responders, defined as a response over the known minimal detectable change or minimal important difference for included tests, will be determined, and compared between HIIT and MICT.
Feasibility of interventions: Completion rate | 12-weeks and 24-months
  Completion rate is determined by the total number of participants still performing the exercise training intervention at 12-week and 24-month follow-up. Reasons for non-completion are also obtained.
Feasibility of interventions: Attendance rate | 12-weeks and 24-months
  Attendance rate is determined by the total number of attended sessions divided by total number of sessions prescribed, presented as a percentage. Reasons for non-attendance are also obtained.
Feasibility of interventions: Exercise fidelity | Throughout the whole intervention period (24-months)
  Exercise fidelity is determined as the incidence of exercise sessions requiring modifications, defined as any deviation from the prescribed exercise.
Feasibility of interventions: Adherence to exercise duration and intensity | Throughout the whole intervention period (24-months)
  Adherence to exercise duration is determined as the adherence to the predefined intervals/minutes of the exercise training. Reasons for non-adherence are also obtained. Adherence to exercise intensity is determined as the adherence to the prescribed intensity of the exercise training. Reasons for non-adherence are also obtained. Exercise intensity (absolute workload [W], relative intensity [% of MAP, % of MPO6], the level of dyspnoea and leg fatigue [0-10, arbitrary units] on the Borg CR10 scale and perceived exertion [6-20, arbitrary units] on the Borg Rating of RPE scale.
Feasibility of interventions: Satisfaction | Throughout the whole intervention period (24-months)
  Participant satisfaction with the performed exercise training (supramaximal HIIT / MICT) will be recorded by adaptation of an existing patient satisfaction questionnaire previously used cycling exercises in COPD. (Evans et. al. Ann Am Thorac Soc 2015)
Feasibility of interventions: Affective responses | Throughout the whole intervention period (24-months)
  Affective response/mood will be measured using the Feeling scale, during and after exercise sessions. The Feeling scale ranges from -5 to +5, where a higher score indicates a better feeling.
Adverse events | Throughout the whole intervention period (24-months)
  Adverse events are rated into four different categories: 1) minor and temporary, 2) serious symptoms (potential risk of severe injury or life threatening, 3) manifest injury or disease, and 4) death, as previously described. An adverse event rate will be calculated for each participant as the total number of sessions during which any adverse events occurred divided by the total number of attended sessions.
Experiences of exercising and its effects | 12 weeks, 24-months
  Face-to-face interviews will explore the participants' experiences and perceptions of participating in the program.
Hospitalisations | 24 months
  Number of hospitalisations per participant during the study period. Time, cause, length of stay, and emergency room visits (with no hospitalization afterwards) and their cause will also be extracted. Hospitalizations and emergency room visits will be classified as respiratory or non-respiratory. In Phase 2, data on hospitalizations will be extracted from the participant's medical record and cross-checked with the participant's diary.
Mortality | 24 months
  Number of deaths during the study period will be extracted from the participant's medical record. Time and cause of each death will also be extracted.
Exacerbations | 24 months
  In the COPD groups, number of exacerbations during the whole study period will be recorded during the whole study period. In Phase 2, data on exacerbations will be extracted from the participant's medical record and cross-checked with the participant's diary.

OTHER OUTCOMES:
Baseline global cognitive function | Baseline
  Baseline global cognitive function, as determined by the Z-score derived from CANTAB and TMT-test battery (primary outcome) will be compared between the groups at baseline to compare the different cohorts (COPD versus healthy controls).
Baseline cardiorespiratory fitness | Baseline
  Baseline cardiorespiratory fitness will be compared between the groups at baseline to compare the different cohorts (COPD versus healthy controls). Measured as maximum oxygen uptake (VO2peak [ml O2/min/kg]) during a standardized ramp-protocol cardiopulmonary exercise test (CPET) on a cycle ergometer.
Baseline muscle power | Baseline
  Baseline cardiorespiratory fitness will be compared between the groups at baseline to compare the different cohorts (COPD versus healthy controls). Peak power (Nm/s) assessed during a seated leg extension in a dymanometer (Biodex System 4).
Baseline brain structure | Baseline
  Baseline brain structured assessed in MRI will be compared between the groups to compare the different cohorts (COPD versus healthy controls). Volume (mm3), area (mm2) and cortical thickness (mm) will be the unit of measure.
Baseline neuroinflammation | Baseline
  Baseline neuroinflammation assessed in PET/CT will be compared between the groups to compare the different cohorts (COPD versus healthy controls). Neuroinflammation is measured as uptake rate (ki) of 11C-deprenyl in the brain assessed
Baseline cognitive function: Montreal Cognitive Assessment (MoCA) | Baseline
  Baseline cognitive function assessed with the MoCA will be investigated at baseline to compare the different cohorts (COPD vs healthy controls) and any differences in cognitive impairment at baseline. The MoCA evaluates multiple domains of cognitive function and yields a score, 0-30 points, where higher is better.
Baseline neurotrophic factors | Baseline
  Neurotrophic factors will be investigated at baseline to compare the different cohorts (COPD versus healhy controls). Levels of BDNF, irisin, IGF-1, Cathepsin B and clusterin in venous blood samples. Unit of measure is pq/ml
Baseline inflammatory markers | Baseline
  Markers of systemic inflammation at baseline will be investigated to compare the different cohorts (COPD versus healthy controls). Levels of interleukin-6, interleukin-8 and TNF-alpha in venous blood, measured in pq/mL, will be assessed.
Baseline chronic inflammation | Baseline
  Baseline chronic inflammation, assessed as hs-CRP (mg/L) will be investigated at baseline to compare the different cohorts (COPD versus healthy controls)
Baseline fibrinogen | Baseline
  Baseline fibrinogen levels (g/L) will be investigated at baseline to compare the different cohorts (COPD versus healthy controls).
Baseline resting lactate | Baseline
  Baseline lactate (mmol/L) will be investigated at baseline to compare the different cohorts (COPD versus healthy controls).
Baseline proportion of slow and fast subtypes of contractile myosin heavy chain isoforms | Baseline
  Proportion of slow and fast subtypes of contractile myosin heavy chain isoforms will be assessed at baseline to compare the different cohorts (COPD versus healthy controls). The tissue sample obtained from the vastus lateralis muscle will be examined with immunohistochemistry techniques to categorize fiber types. Expressed as relative distribution in percent and relative area of the muscle in percent.
Baseline mitochondrial biogenesis | Baseline
  mRNA and protein levels of peroxisome proliferator-activated receptor gamma coactivator 1 (PGC-1) alpha and PGC-1beta will be investigated at baseline to compare the different cohorts (COPD versus healthy controls). Unit of measure is fold-change or arbitrary units.
Baseline enzyme content | Baseline
  Enzyme content will be investigated at baseline to compare the different cohorts (COPD versus healthy controls). Including phosphofructokinase (PFK; glycolysis), lactate dehydrogenase (LDH; anaerobic glycolysis), citrate synthase (CS; Krebs cycle), succinate dehydrogenase (SDH; Krebs cycle), 3-hydroxyacyl Coenzyme A dehydrogenase (HADH; beta-oxidation) and mitochondrial complex I-V. Unit of measure is micromol/min/g tissue.

CONTACTS AND LOCATIONS:
Overall Officials: André Nyberg, PhD, Principal Investigator — Umeå University
Locations (2):
- Hasselt University, Hasselt, Diepenbeek, Belgium
- Umeå University, Umeå, Sweden

IPD SHARING:
Plan to Share IPD: Yes
We strive to share all the IPD that underlie results in a publication in a open data repository, if this will be possible given regulations and agreements at that time.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: IPD will become available 6 months after publication. The full study protocol including the analysis plan will be submitted for publication during 2023. Informed consent forms and other supporting material will be available on a reasonable request to the principal investigator.
Access Criteria: The principal investigator will review requests for supporting material. IPD will be open access in a data repository.

REFERENCES:
- [Derived] Jakobsson J, Burtin C, Hedlund M, Boraxbekk CJ, Westman J, Karalija N, Stal P, Sandstrom T, Ruttens D, Gosker HR, De Brandt J, Nyberg A. Effects and mechanisms of supramaximal high-intensity interval training on extrapulmonary manifestations in people with and without chronic obstructive pulmonary disease (COPD-HIIT): study protocol for a multi-centre, randomized controlled trial. Trials. 2024 Oct 8;25(1):664. doi: 10.1186/s13063-024-08481-3. PMID 39375781
- See also: Study site at Umeå University — https://www.umu.se/en/research/projects/copd-hiit/